CLINICAL TRIAL: NCT06867016
Title: Effects of Bidomain Cognitive and Aerobic Training on Cognitive Functioning in Mild Cognitive Impairment.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/MS-PT/O2029 Saliha Ashfaq
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognition; Old age; mild cognitive impairment; aerobic; cognitive training
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Cognitive & Aerobic Training Group (Experimental): The ACT combined training will consist of simultaneous aerobic exercise and cognitive training in a dual-task format.
  Interventions: Other: Combined Cognitive & Aerobics Training
- Cognitive Training Group (Active Comparator): Cognitive training group include cognitive training involving speed processing, memory recall, problem-solving, and visual attention exercises.
  Interventions: Other: Cognitive Training

INTERVENTIONS:
Other: Combined Cognitive & Aerobics Training — The ACT combined training will consist of simultaneous aerobic exercise and cognitive training in a dual-task format, conducted twice a week for 8 weeks. The aerobic training (AT) will consist of twice-weekly sessions that include yoga, brisk walking, pedaling exercises, and step aerobics, alongside cognitive training involving speed processing, memory recall, problem-solving, and visual attention exercises. Each session will last approximately 20 minutes, and assessments will be performed at baseline, 4th week, and 8th week.
  Arms: Combined Cognitive & Aerobic Training Group
Other: Cognitive Training — Cognitive training involving speed processing, memory recall, problem-solving, and visual attention exercises. Each session will last approximately 20 minutes, and assessments will be performed at baseline, the 4th week, and the 8th week.
  Arms: Cognitive Training Group

SUMMARY:
The study aims to assess the effects of Bidomain cognitive and aerobic training on both cognitive functioning and quality of life in individuals with mild cognitive impairment.

DETAILED DESCRIPTION:
The proposed study addresses a notable gap in the literature regarding the comparison between combined cognitive-aerobic training and cognitive training alone in improving cognitive function for patients with mild cognitive impairment (MCI). While previous studies have demonstrated the positive effects of both training methods on cognitive function independently, there is currently no research directly comparing their effectiveness when used together. The study aims to provide evidence on which treatment regime-combined cognitive-aerobic training or cognitive training alone-offers better outcomes for MCI patients. Aerobic training is known to enhance brain structure and function by strengthening neuronal connections, largely due to increased levels of brain-derived neurotrophic factor (BDNF) and enhanced vascularization, which stimulates hippocampal growth. On the other hand, cognitive training improves global cerebral functional connectivity, particularly activating the prefrontal cortex, which leads to better cognitive performance. Combining these training modalities may yield greater benefits than focusing on just one, offering a cost-effective, accessible approach that could significantly improve the quality of life and daily functioning for individuals with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Older adults 60 years & above
* With normal vision and color perception
* Independent Individual capable of carrying out daily tasks
* Individuals scoring 21-25 on the Mini-Mental State Examination (MMSE)

Exclusion Criteria:

* Medication affecting the exercise capacity of individual
* Regular participation in aerobic training for the last six months
* Cardiovascular or other diseases that do not allow physical activity
* A diagnosed severe psychiatric disease (e.g., depression)
* Patients with cognitive impairment or other neurological impairments due to AD or dementia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-08-28 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Mini-mental state examination (MMSE) | 8 weeks
  The Mini-Mental State Examination (MMSE) is a widely used screening test for cognitive deficits, with scores ranging from 0 to 30. A score of 24 or below indicates potential cognitive impairment, particularly for patients aged 65 and older. The MMSE evaluates verbal abilities, where scores of 30-27 are considered normal, while lower scores indicate mild (26-21 points), moderate (20-10 points), or severe (9-0 points) dementia.
Short Cognitive Test (SKT) | 8 weeks
  The SKT (Syndrom-Kurz-Test) is a recognized short cognitive performance test used to detect attention and memory deficits. It features subtest norm values ranging from 0 to 3, with a total score ranging from 0 to 27, where higher scores indicate more severe cognitive impairment. The SKT assesses memory performance and attention based on processing speed.
  The SKT (Syndrom-Kurz-Test) is a recognized short cognitive performance test used to detect attention and memory deficits. It features subtest norm values ranging from 0 to 3, with a total score ranging from 0 to 27, where higher scores indicate more severe cognitive impairment. The SKT assesses memory performance and attention based on processing speed.

SECONDARY OUTCOMES:
World health observational quality of life-BREF-100 | 8 weeks
  Quality of life (QOL) is essential for understanding the subjective experience of mild cognitive impairment (MCI) and its impact on individuals. In the WHOQOL-BREF questionnaire, scores range from 0 (worst possible health) to 100 (best possible health), with higher scores indicating better QOL. Each domain score is calculated by taking the mean of items within that domain and then transformed linearly to a 0-100 scale

CONTACTS AND LOCATIONS:
Overall Officials: Saliha Ashfaq, MS-NMPT*, Principal Investigator — Riphah International University
Locations (1):
- DHQ Chakwal, Chakwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No